CLINICAL TRIAL: NCT06649448
Title: A Multi-cohort, Open-label, Multi-center Exploratory Study of Efbemalenograstim Alfa Injection for Preventing Absolute Neutrophil Count (ANC) Reduction in Solid Tumor Patients Undergoing Immune-chemotherapy Regimen.
Brief Title: A Multi-cohort Study of Efbemalenograstim Alfa Injection for Preventing ANC Reduction in Solid Tumor Patients Post Immune-chemotherapy.
Acronym: EF-001
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Investigator Official Title President of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDZLEC2024-115-02
Record Dates: First submitted 2024-10-09; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor Cancer; Chemotherapy Induced Neutropenia; G-CSF
Keywords: ICI combined with chemotherapy; ANC; G-CSF; Solid Tumor
MeSH Terms: interventions — Carboplatin; PE regimen; Paclitaxel; Cisplatin; Pemetrexed; TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Small cell lung cancer (SCLC) patients receiving ICI combined with chemotherapy (etoposide + carboplatin/cisplatin).
  Interventions: Drug: Efbemalenograstim alfa Injection; Drug: carboplatin/cisplatin-etoposide
- Cohort 2 (Experimental): Non-small cell lung cancer (NSCLC) patients receiving ICI combined with chemotherapy (platinum-based/taxane, pemetrexed/platinum).
  Interventions: Drug: Efbemalenograstim alfa Injection; Drug: Carboplatin plus Paclitaxel; Drug: Cisplatin/pemetrexed or Carboplatin/pemetrexed
- Cohort 3 (Experimental): Esophageal squamous cell carcinoma (ESCC) patients receiving ICI combined with chemotherapy (TP, which stands for cisplatin + taxane).
  Interventions: Drug: Efbemalenograstim alfa Injection; Drug: TP regimen

INTERVENTIONS:
Drug: Efbemalenograstim alfa Injection — This product should be administered subcutaneously 48 hours after the completion of anti-tumor drug administration in each chemotherapy cycle. The recommended dose for adults is 20mg administered subcutaneously once per chemotherapy cycle. Please do not administer this product within 14 days before and 24 hours after the administration of cytotoxic chemotherapy drugs.
Drug: carboplatin/cisplatin-etoposide — one of the following chemotherapy regimens can be selected: EC, Q3W: Carboplatin AUC = 5~6 on Day 1; Etoposide 80~100 mg/m² on Days 1-3. EP, Q3W: Cisplatin 75~80 mg/m² on Day 1; Etoposide 80~100 mg/m² on Days 1-3.
  Arms: Cohort 1
Drug: Carboplatin plus Paclitaxel — For non-small cell lung cancer (squamous cell carcinoma), one of the following chemotherapy regimens can be selected:
  Carboplatin AUC = 5~6 on Day 1 + Taxane: Paclitaxel 175-200 mg/m² on Day 1; or Albumin-bound Paclitaxel 200-260 mg/m² on Day 1, administered every 3 weeks (Q3W); Cisplatin/Carboplatin 75 mg/m²/AUC = 5~6 on Day 1 + Gemcitabine 1000 mg/m² on Days 1 and 8, administered every 3 weeks (Q3W).
  Arms: Cohort 2
Drug: Cisplatin/pemetrexed or Carboplatin/pemetrexed — For non-small cell lung cancer (non-squamous cell carcinoma), one of the following chemotherapy regimens can be selected:
  Cisplatin 75 mg/m² on Day 1 + Pemetrexed 500 mg/m² on Day 1, administered every 3 weeks (Q3W).
  Carboplatin AUC = 5~6 on Day 1 + Pemetrexed 500 mg/m² on Day 1, administered every 3 weeks (Q3W).
  Arms: Cohort 2
Drug: TP regimen — The chemotherapy regimen options include:
  TP regimen: Cisplatin 60-80 mg/m² administered via intravenous drip on Day 1 + Taxane: Paclitaxel 175 mg/m² on Day 1; or Albumin-bound Paclitaxel 200-260 mg/m² on Day 1, with a treatment cycle of every 3 weeks (Q3W).
  Arms: Cohort 3

SUMMARY:
This study is a multi-cohort, open-label, multi-center exploratory clinical research designed to evaluate the efficacy and safety of Efbemalenograstim alfa Injection in preventing neutropenia (reduction in absolute neutrophil count, ANC) in solid tumor patients undergoing immune checkpoint inhibitor (ICI) combined chemotherapy. A total of 200 solid tumor patients who are scheduled to receive at least 2 cycles of ICI combined chemotherapy will be enrolled. The study is divided into three cohorts:

Cohort 1: Small cell lung cancer (SCLC) patients receiving ICI combined with chemotherapy (etoposide + carboplatin/cisplatin).

Cohort 2: Non-small cell lung cancer (NSCLC) patients receiving ICI combined with chemotherapy (platinum-based/taxane, pemetrexed/platinum).

Cohort 3: Esophageal squamous cell carcinoma (ESCC) patients receiving ICI combined with chemotherapy (TP, which stands for cisplatin + taxane).

DETAILED DESCRIPTION:
This study is a multi-cohort, open-label, multi-center exploratory clinical trial aimed at evaluating the efficacy and safety of Efbemalenograstim alfa Injection in preventing neutropenia (reduction in absolute neutrophil count, ANC) in solid tumor patients undergoing immune checkpoint inhibitor (ICI) combined chemotherapy. It plans to enroll 200 solid tumor patients who are scheduled to receive at least 2 cycles of ICI combined chemotherapy. The study is divided into three cohorts:

Cohort 1: Small cell lung cancer (SCLC) patients receiving ICI combined with chemotherapy (etoposide + carboplatin/cisplatin).

Cohort 2: Non-small cell lung cancer (NSCLC) patients receiving ICI combined with chemotherapy (platinum-based/taxane, pemetrexed/platinum).

Cohort 3: Esophageal squamous cell carcinoma (ESCC) patients receiving ICI combined with chemotherapy (TP, which stands for cisplatin + taxane).

Eligible patients will receive Efbemalenograstim alfa Injection (20 mg/dose, subcutaneous injection) 24-72 hours after the end of each chemotherapy cycle, from the 1st to the 4th cycle of ICI combined chemotherapy. Investigators must ensure that the first cycle of chemotherapy is administered at the recommended dose according to the protocol. For the 2nd to 4th cycles, dose delays or adjustments due to toxicity are allowed, and investigators may also determine the individual chemotherapy cycles and drug doses based on the patient's specific condition during these cycles. After completing 4 cycles of ICI combined chemotherapy and evaluation, patients will receive subsequent treatment according to standard clinical practice.

Referencing the 2023 CSCO Guidelines, the recommended ICI combined chemotherapy regimens for subjects are as follows:

Cohort 1 - SCLC, referring to the "2023 CSCO Guidelines for the Diagnosis and Treatment of SCLC":

Immune drugs (choose one):

Atezolizumab 1200 mg, d1, Q3W Durvalumab 1500 mg, d1, Q3W Serplulimab 4.5 mg/kg, d1, Q3W Adebelimab 20 mg/kg, d1, Q3W

Chemotherapy regimens (choose one):

EC, Q3W: Carboplatin AUC=5-6, d1; Etoposide 80-100 mg/m2, d1-3 EP, Q3W: Cisplatin 75-80 mg/m2, d1; Etoposide 80-100 mg/m2, d1-3

Cohort 2 - NSCLC, referring to the "2023 CSCO Guidelines for the Diagnosis and Treatment of NSCLC":

NSCLC (Squamous Cell Carcinoma) - Immune drugs (choose one):

Pembrolizumab 200 mg, d1, Q3W Camrelizumab 200 mg, d1, Q3W Sintilimab 200 mg, d1, Q3W Tislelizumab 200 mg, d1, Q3W Serplulimab 4.5 mg/kg, d1, Q3W Atezolizumab 1200 mg, d1 + Bevacizumab 15 mg/kg, d1, Q3W Sugemalimab 1200 mg, d1, Q3W Anplitumab 200 mg, d1, Q3W

NSCLC (Squamous Cell Carcinoma) - Chemotherapy regimens (choose one):

Carboplatin AUC=5-6, d1 + Taxane: Paclitaxel 175-200 mg/m2, d1; or Albumin-bound Paclitaxel 200-260 mg/m2, d1, Q3W Cisplatin/Carboplatin 75 mg/m2/AUC=5-6, d1 + Gemcitabine 1000 mg/m2, d1, d8, Q3W

NSCLC (Non-Squamous Cell Carcinoma) - Immune drugs (choose one):

Pembrolizumab 200 mg, d1, Q3W Camrelizumab 200 mg, d1, Q3W Sintilimab 200 mg, d1, Q3W Tislelizumab 200 mg, d1, Q3W Atezolizumab 1200 mg, d1 Sugemalimab 1200 mg, d1, Q3W

NSCLC (Non-Squamous Cell Carcinoma) - Chemotherapy regimens (choose one):

Cisplatin 75 mg/m2, d1 + Pemetrexed 500 mg/m2, d1, Q3W Carboplatin AUC=5-6, d1 + Pemetrexed 500 mg/m2, d1, Q3W

Cohort 3 - ESCC, referring to the "2023 CSCO Guidelines for the Diagnosis and Treatment of Esophageal Cancer":

Immune drugs (choose one):

Camrelizumab 200 mg, d1, Q3W Toripalimab 240 mg, d1, Q3W Sintilimab 200 mg, d1, Q3W Tislelizumab 200 mg, d1, Q3W Serplulimab 3 mg/kg intravenous infusion, d1, Q2W

Chemotherapy regimen:

TP regimen: Cisplatin 60-80 mg/m2 intravenous infusion, d1 + Taxane: Paclitaxel 175 mg/m2, d1; or Albumin-bound Paclitaxel 200-260 mg/m2, d1, Q3W Note: The chemotherapy schedule for cisplatin and etoposide can be modified as needed, while maintaining the total dose administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-ups;
* Aged 18 years or older, regardless of gender;
* Patients with histologically or cytologically confirmed stage IV small cell lung cancer (SCLC) (as per the 8th edition of the American Joint Committee on Cancer (AJCC)) or T3-4 SCLC with multiple pulmonary nodules or tumors/nodules too large to be included in a tolerable radiotherapy plan, stage IV non-small cell lung cancer (NSCLC) (as per the 8th edition of the International Association for the Study of Lung Cancer (IASLC) Thoracic Oncology Staging Manual), or stage IV esophageal squamous cell carcinoma (excluding adenosquamous carcinoma) who are not eligible for radical therapy;
* Patients who have not previously received systemic anti-tumor therapy for advanced/metastatic disease. For patients who have received neoadjuvant/adjuvant and radical concurrent chemoradiotherapy, screening is allowed if the time from the last chemotherapy to recurrence or progression exceeds 6 months. For patients who have received radiotherapy alone, screening is allowed after disease progression;
* Patients planned to receive immunotherapy combined with at least 2 cycles of chemotherapy regimens with a high risk of severe neutropenia complicated by febrile neutropenia (FN) or medium FN risk regimens combined with ≥ 1 patient-specific risk factor. According to the "Chinese Expert Consensus on Diagnosis and Treatment of Neutropenia Induced by Chemotherapy for Cancer (2023 Version)", patient-specific factors are also crucial in influencing the risk of FN. The patient factors that increase the risk of FN mainly include: (1) Age > 65 years and receiving full-dose chemotherapy; (2) Prior chemotherapy or radiotherapy; (3) Persistent neutropenia (>10 days); (4) Bone marrow invasion by tumor; (5) Recent surgery and/or open trauma; (6) Poor overall physical condition with comorbidities such as liver (serum bilirubin > 2 times the upper limit of normal (ULN)), kidney (creatinine clearance ≤ 50 ml/min), heart, lung, endocrine, and other underlying diseases; (7) Poor nutritional status; (8) Chronic immunosuppression, such as human immunodeficiency virus infection, organ transplantation, and long-term immunosuppression after transplantation; (9) Advanced disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score: 0-1;
* Adequate organ and bone marrow function:

  1. Blood routine examination criteria (without blood transfusion or blood products and without using G-CSF or other hematopoietic stimulating factors within 14 days to correct):

     Hemoglobin (HB) ≥ 80g/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet count (PLT) ≥ 100×109/L;
  2. Biochemical examination criteria:

     Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5´ ULN; if there is liver metastasis, then ALT and AST ≤ 5´ ULN; Serum creatinine ≤ 1.5´ ULN;
  3. Left ventricular ejection fraction > 50%;
* The investigator judges that the patient can tolerate the treatment with Abegrimacostat Alpha.

Exclusion Criteria:

* Patients diagnosed with acute congestive heart failure, cardiomyopathy, or myocardial infarction through clinical examination, electrocardiogram, or other means;
* Individuals with a history of rubber allergy;
* Patients who have received radiotherapy for bone lesions (patients who have received radiotherapy for lesions other than bone lesions can be enrolled 4 weeks after treatment);
* Patients who have undergone bone marrow transplantation or stem cell transplantation;
* Pregnant or lactating women;
* Patients with alcoholism or drug abuse that affects their compliance in participating in the study;
* Known allergy to granulocyte colony-stimulating factors or excipients in the study drug;
* Use of other investigational drugs within 1 month prior to enrollment in this study;
* Received treatment with recombinant human granulocyte colony-stimulating factor within 6 weeks prior to enrollment;
* Presence of other primary malignancies, with the following exceptions: 1) Malignancies in complete remission for at least 2 years prior to enrollment and requiring no additional treatment during the study; 2) Non-melanoma skin cancer or malignant lentigo maligna that has been adequately treated and shows no evidence of disease recurrence; 3) Carcinoma in situ that has been adequately treated and shows no evidence of disease recurrence;
* The investigator believes that the patient has a disease or symptom that makes them unsuitable for participation in this study, or that the study drug may harm the patient's health or affect the assessment of adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of ≥ Grade 3 neutropenia in the first chemotherapy cycle | At the end of Cycle 1 (each cycle being 21 days)
  The incidence rate of ≥ Grade 3 neutropenia in the first chemotherapy cycle, defined as the percentage of individuals with ANC < 1.0×109/L in the first chemotherapy cycle among the analyzed population.

SECONDARY OUTCOMES:
The incidence rate of ≥ Grade 3 neutropenia in the second and subsequent cycles | At the end of the second and subsequent chemotherapy cycles(each cycle being 21 days)
  The incidence rate of ≥ Grade 3 neutropenia in the second and subsequent cycles, defined as the percentage of individuals with ANC < 1.0×109/L in chemotherapy cycles 2-4 among the analyzed population;
The nadir (lowest value) of neutrophils in the first cycle | At the end of Cycle 1 (each cycle being 21 days)
  The nadir (lowest value) of neutrophils in the first cycle, defined as the lowest count (trough value) of neutrophils in the first cycle;
The time required for the nadir of neutrophils to recover above 2×109/L in each cycle | From the start of treatment to the end of treatment
  The time required for the nadir of neutrophils to recover above 2×109/L in each cycle, defined as the time (in days) required for the ANC nadir to recover above 2×109/L in each cycle.
The incidence rate and duration of FN (Febrile Neutropenia) in each cycle | From the start of treatment to the end of treatment
  The incidence rate and duration of FN (Febrile Neutropenia) in each cycle, defined as the percentage of individuals experiencing FN [oral temperature > 38.3°C or oral temperature > 38.0°C measured twice consecutively within 2 hours, with ANC < 0.5×109/L or predicted to be < 0.5×109/L] [23] among the analyzed population, and the duration (in days) of FN episodes;
The duration of ≥ Grade 3 neutropenia in each cycle | From the start of treatment to the end of treatment
  The duration of ≥ Grade 3 neutropenia in each cycle, defined as the duration (in days) of ANC < 1.0×109/L in each cycle;

CONTACTS AND LOCATIONS:
Overall Officials: JinMing Yu, Phd, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided